CLINICAL TRIAL: NCT05312749
Title: The Effect of Web-Based Progressive Muscle Relaxation Exercise on the Perceived Stress and Anxiety Level of Nursing Students Found in Clinical Practice for the First Time: A Randomized Controlled Trial
Brief Title: The Effect of Web Based Progressive Muscle Relaxation Exercise on Clinical Stress and Anxiety of Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, gülcan bahcecioğlu, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2021/09-45
Record Dates: First submitted 2022-03-16; First posted 2022-04-05 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Anxiety; Stress; Nursing Students; Relaxation Program
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: (Experimental): Experimental: will do progressive relaxation exercises
  Interventions: Other: progressive relaxation exercises
- Control (No Intervention): won't do progressive relaxation exercises

INTERVENTIONS:
Other: progressive relaxation exercises — progressive relaxation exercises
  Other Names: progressive muscle relaxation exercises
  Arms: Experimental:

SUMMARY:
Purpose: The study was conducted to examine the effect of web-based progressive muscle relaxation exercise on the perceived stress and anxiety level of nursing students who were in clinical practice for the first time.

Method: This randomized controlled study was conducted at a state university in Turkey. The sample of the study consisted of a total of 66 nursing students, 36 of whom were control and 30 interventions, who were educated in the 2021-2022 academic year, were in clinical practice for the first time and agreed to participate in the research. The intervention group was asked to perform a total of 36 sessions of progressive muscle relaxation exercise, 3 days a week for 12 weeks. Data; It was collected using the "Sociodemographic Characteristics Form", "State-Trait Anxiety Inventory (DSQ)" and "Perceived Stress Inventory (PSI)".

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old
* Studying in the 2021-2022 academic year
* Being in 2nd grade
* Not going into clinical practice before

Exclusion Criteria:

* Being under the age of 18
* Not studying in the 2021-2022 academic year
* Being in 1st, 3rd or 4th grade
* Prior clinical practice

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2021-12-25 (Actual)

PRIMARY OUTCOMES:
The State-Trait Anxiety Inventory | 12 week
  The State-Trait Anxiety Inventory was developed by Spielberger et al. (1970) (Spielger, Gorsuch, & Lushene, 1970). The validity and reliability of the scale in Turkey was established by Öner and Le Compte (1983) (Öner & Le Compte, 1983). The scale consists of two parts, the State Anxiety Inventory and the Trait Anxiety Inventory. The first 20 items assess situational anxiety, and the last 20 items assess trait anxiety. In this study, the "State Anxiety Inventory", which is the first 20 items, was used to evaluate situational anxiety. State Anxiety Scale; It was developed to determine how an individual feels at a certain moment and under certain conditions. The scale is 4-point Likert type. Scores from the scale range from 20 to 80. Higher scores indicate higher levels of anxiety.
Perceived Stress Scale | 12 week
  The Perceived Stress Scale was developed by Cohen, Kamarck, and Mermelstein in 1983 to determine the level of stress that threatens human health (Cohen et al. 1983). Its Turkish validity and reliability were determined by Eskin et al. (2013) (Eskin et al., 2013). PSS-14 consists of 2 factors: "insufficient self-efficacy" and "stress" perception. The scale is a 5-point Likert type scale and consists of 14 items. As the scores obtained from the scale increase, the level of stress perceived by the person also increases. PSS scores range from 0 to 56, with 0-35 point range indicating normal stress level and 35-56 point range indicating that the individual is under stress.

CONTACTS AND LOCATIONS:
Overall Officials: Gülcan B.TURAN, PH, Study Director — Firat University
Locations (2):
- Turkey (Türkiye) (2):
  - Atatürk university nursing faculty, Erzurum, Center
  - Fırat Üniversitesi, Elâzığ

IPD SHARING:
Plan to Share IPD: No
The article is intended to be shared after it is published.